CLINICAL TRIAL: NCT03110783
Title: A Prospective, Randomized, Controlled, Single Blinded, Study to Evaluate the Safety and Effectiveness of Bioseal as an Adjunct to Sutured Dural Repair
Brief Title: Bioseal Dural Sealing Study BIOS-14-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou Bioseal Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOS-14-001
Record Dates: First submitted 2017-03-22; First posted 2017-04-12 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Benign Tumors; Malignant Tumors; Vascular Malformation
Keywords: Bioseal as an Adjunct to Sutured Dural Repair; elective posterior fossa; supratentorial procedure
MeSH Terms: conditions — Neoplasms; Vascular Malformations | interventions — Bioseal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- suture (control) (No Intervention): Subjects randomized to control will receive additional dural sutures as deemed necessary by the surgeon. CSF leakage will be re-evaluated with the Valsalva maneuver to 10-20 cm H2O for 5 to 10 seconds. Closure of the remaining layers of the surgical site will be performed according to the surgeon's standard of practice.
- Bioseal (Experimental): Subjects randomized to receive Bioseal, a thin layer will be applied to the entire length of the suture line and the adjacent area to approximately 5mm away, including all suture holes. Up to two layers of Bioseal may be used for each application. While Bioseal achieves complete coagulation, CSF leakage will be re-evaluated with the Valsalva maneuver to 10-20 cm H2O for 5 to 10 seconds. Up to two applications (one application includes applying up to two layers of Bioseal product followed by the CSF leakage re-evaluation with Valsalva maneuver) per subject are allowed. Closure of the remaining layers of the surgical site will be performed according to the surgeon's standard of practice.
  Interventions: Biological: Bioseal

INTERVENTIONS:
Biological: Bioseal — Upon completion of the sutured dural repair, the closure will be evaluated for intra-operative CSF leakage with a baseline Valsalva maneuver to 10-20 cm H2O for 5-10 seconds. Subjects who have a CSF leak will be enrolled into the study. If randomized to receive Bioseal, a thin layer will be applied to the entire length of the suture line and the adjacent area to approximately 5mm away, including all suture holes. Up to two layers of Bioseal may be used for each application. While Bioseal achieves complete coagulation, CSF leakage will be re-evaluated with the Valsalva maneuver to 10-20 cm H2O for 5 to 10 seconds.
  Arms: Bioseal

SUMMARY:
A Prospective, Randomized, Controlled, Single Blinded, Study to Evaluate the Safety and Effectiveness of Bioseal as an Adjunct to Sutured Dural Repair

DETAILED DESCRIPTION:
This is a randomized, single blinded, multi-center controlled study evaluating the effectiveness of Bioseal as an adjunct to sutured dural closure compared to control to obtain an intra-operative watertight dural closure.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative

  1. Patient undergoing elective craniotomy/craniectomy for pathological processes (such as benign and malignant tumors, vascular malformation) in the posterior fossa or in the supratentorial region.
  2. Age ≥ 18 years.
  3. Patients who are able and willing to comply with the procedures required by the protocol.
  4. Signed and dated written informed consent from the subject or from his/her legal representative prior to any study-specific procedures.
* Intraoperative

  1. Patient undergoing elective craniotomy/craniectomy for pathological processes (such as benign and malignant tumors, vascular malformation) in the posterior fossa or in the supratentorial region and who are demonstrated to have persistent CSF leakage following suture closure of the dural incision. CSF leakage will be evaluated during a period of Valsalva of 10-20 cm of H20 for 5-10 seconds. If a spontaneous leak is apparent immediately after dural closure, no Valsalva will be performed.
  2. Surgical wound classification Class I. Penetration of mastoid air cells during partial mastoidectomy is permitted.
  3. The cuff of native dura along the craniotomy edge is ≥10 mm wide, to facilitate suturing and to allow for sufficient surface area for adherence of the investigational product.

Exclusion Criteria:

* Preoperative

  1. Subjects with a dura lesion from a recent surgery that still has the potential for CSF leakage.
  2. The previous craniotomy/ craniectomy within 6 months or radiation therapy within 2 years before this surgery.
  3. Chemotherapy or radiation therapy scheduled within 7 days following surgery.
  4. Subjects with severely altered renal (serum creatinine >2 mg/dL) and/or hepatic function [ALT, AST > 5 x upper limit of norm (ULN)].
  5. Severe Anemia (Hemoglobin <60 g/L) or Hypoproteinemia (Total protein <60 g/L or 6g% ) .
  6. Non-compliant or insufficient treatment of diabetes mellitus [glycosylated hemoglobin (HbA1c) > 7.5%].
  7. Conditions compromising the immune system; existence of autoimmune disease.
  8. Evidence of a potential infection: fever >38℃, WBC <3500/uL or >13000/uL, positive urine culture, positive blood culture, positive chest X-ray, evidence of infection along the planned surgical path.
  9. Known hypersensitivity to the porcine fibrin sealant product.
  10. Female subjects of childbearing potential with a positive urine or serum pregnancy test within 7 days prior to surgery.
  11. Female subjects who are breastfeeding or intend to become pregnant during the clinical study period.
  12. Participation in another clinical trial with exposure to another investigational drug or device within 30 days prior to enrolment.
* Intraoperative

  1. Native dura cuff during craniotomy/craniectomy that cannot be completely repaired.
  2. Use of implants made of synthetic materials coming into direct contact with dura (e.g., PTFE patches, shunts, ventricular and subdural drains).
  3. Occlusive hydrocephalus caused by posterior fossa pathology or partial blockage of CSF pathways during surgical procedure.
  4. Existing CSF drains on the surgical path.
  5. Use of other fibrin sealants for hemostasis.
  6. Placement of Gliadel Wafers or similar products.
  7. Persistently increased brain surface tension that may lead to an incomplete repair requiring.
  8. Intersecting durotomy scars in the surgical path from a previous operation that cannot be completely removed by the planned dura resection.
  9. Two or more separate dura defects during surgery.
  10. Others in addition to above exclusion criteria, the subject, in the opinion of the investigator, would not be suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of success (watertight closure) CSF leakage | 5 to 10 seconds after final Valsalva maneuver
  no CSF leakage from dural repair intra-operatively

SECONDARY OUTCOMES:
Incidence of CSF leakage | Up to Discharge, an average of 3-5days in general
  Incidence of CSF leakage post-surgery to discharge
Incidence of CSF leakage | Up to 30(+/-7)Days
  Incidence of CSF leakage 30 (±7) days post operatively
Incidence of adverse events | Up to 30(±7)Days
  Incidence of adverse events
Incidence of surgical site infections (SSI) | Up to 30(± 7) days
  Incidence of surgical site infections (SSI) according to Surgical Site Infection Infection Prevention and Control Guideline (MOH) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ying Mao, MD, PhD, Principal Investigator — Hua Shan Hospital, Shanghai Medical College, Fudan University; Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (10):
- China (10):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The first Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - TongJi Hospital, TongJi Medical College of HUST, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Du S, Zhao J, Qiao G, Wu S, Han Y. Cost-Effectiveness Analysis of the Application of a Porcine-Derived Fibrin Sealant for the Treatment of Cerebrospinal Fluid Leak in China. Clin Ther. 2022 Apr;44(4):575-584. doi: 10.1016/j.clinthera.2022.02.010. Epub 2022 Apr 19. PMID 35450755